CLINICAL TRIAL: NCT06148428
Title: Anxiety-related Fixation Instability During Laser in Situ Keratomileusis (LASIK)
Brief Title: Anxiety-related Fixation Instability During LASIK
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Other Study IDs: ARFILASIK
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Refractive Errors
Keywords: Laser in Situ Keratomileusis; Anxiety; Eye-tracker; Fixation instability
MeSH Terms: conditions — Refractive Errors; Anxiety Disorders | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal group: Based on the Hospital Anxiety and Depression scale anxiety sub-score (HADS anxiety sub-score, the seven-item anxiety sub-score for scaling a patient's anxiety levels before LASIK)
  Patients who had a sub-score of ≤7 denotes no anxiety scale (normal).
  Interventions: Procedure: Laser in situ keratomileusis (LASIK)
- Borderline anxiety group: Based on the Hospital Anxiety and Depression scale anxiety sub-score (HADS anxiety sub-score, the seven-item anxiety sub-score for scaling a patient's anxiety levels before LASIK)
  Patients who had a sub-score of 8-10 denotes doubtful anxiety scale (borderline).
  Interventions: Procedure: Laser in situ keratomileusis (LASIK)
- Anxious group: Based on the Hospital Anxiety and Depression scale anxiety sub-score (HADS anxiety sub-score, the seven-item anxiety sub-score for scaling a patient's anxiety levels before LASIK)
  Patients who had a sub-score of 11-21 is abnormal and denotes a definite anxiety scale (case).
  Interventions: Procedure: Laser in situ keratomileusis (LASIK)

INTERVENTIONS:
Procedure: Laser in situ keratomileusis (LASIK) — Patients were planned to undergo laser in situ keratomileusis. Local anesthesia was achieved by preservative-free oxybuprocaine hydrochloride 0.4% drops (a commonly used topical anesthetic due to its effectiveness in alleviating pain and ocular surface discomfort during the procedure). During surgery, the lights of the operating room were dimmed as much as possible and the surgeons spoke to the patients in a calm voice and explained what was happening. They also reassured the patients that the surgery was going as planned and would be over soon.
  For patients undergoing (Microkeratome) MK-LASIK, a Moria 2 Microkeratome (Moria SA, Antony, France) was used to create the flap. For patients undergoing Femtosecond LASIK (FS-LASIK), the Allegretto Wave Light FS-200 femtosecond Laser (Alcon labs, Fort Worth, TX, USA) was used for flap creation.
  Laser ablation was performed using WaveLight EX500 Excimer Laser (Alcon labs, Fort Worth, TX, USA) with a planned post-operative emmetropia.

SUMMARY:
Anxiety is common among patients undergoing eye surgery, which is typically performed under topical anesthesia while the patient is awake. This can be an unsettling experience for patients, who may worry about being able to keep their eyes still during surgery, cooperate with the surgical team, and remain immobile in an unfamiliar environment. Patients may also experience anxiety due to concerns about surgical pain, possible complications, and the uncertainty of the outcome of the surgery.

In this study, the investigators aimed to investigate the correlation between the severity of anxiety symptoms during LASIK, and fixation instability during photo-ablation as plotted by the eye tracker.

DETAILED DESCRIPTION:
Patient cooperation during LASIK is essential for the surgeon's comfort and predictable results. Fixation instability, which is the inability of the patient to keep their eye still during surgery, is a common problem during LASIK surgery and may lead to unexpected outcomes.

Eye movements occur continually during the excimer ablation. These eye movements can have a large amplitude, a frequency of over 100 Hz, and a corneal speed of around 150 mm/s. With the advancement of scanning-spot excimer lasers, much work has focused on increasing the efficacy of the photo-ablation and smoothness of the ablated surface, especially with respect to the position of the patient's eye by developing state-of-the-art eye trackers to help maintain alignment during photoablation, which can improve refractive outcome.

ELIGIBILITY:
Inclusion Criteria:

* Candidates undergoing LASIK with

  1. Myopia up to 12 diopters
  2. Hyperopia up to 6 diopters
  3. Astigmatism up to 6 diopters

Exclusion Criteria:

1. Previous corneal surgery,
2. Pregnant or lactating females,
3. Concomitant ocular or systemic disease that contraindicated LASIK,
4. Patients with communication barriers, hypochondria, previous stressful surgical experiences, taking psychotropic drugs, or having a history of any clinically relevant psychiatric or cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cohort study was conducted at 2 refractive surgery centers in Assiut city, Egypt (Private practice) and included patients who were candidates for LASIK eye surgery for correction of their refractive errors including myopia, hyperopia and astigmatism.
Sampling Method: Probability Sample
Enrollment: 2435 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
The eye-tracking pupil position plot | Immediately following surgery
  This is a scheme that allows the system to capture the image, process it, and then verify eye position with the next image before releasing the pulse. After treatment, the system releases a summarized treatment report including a plot that depicts various pupil center positions within 3.0 mm off-center (on x and y axes) relative to the eye tracking cameras during ablation.

SECONDARY OUTCOMES:
Heart rate | During and at the end of surgery.
  Upon entering the operating room, patients were attached to a pulse oximeter, and an operating room nurse recorded the heart rate (HR) at the start of the operation, during flap creation, during ablation, and at the end of surgery.
Subjective evaluation of patient's cooperation by surgeon: | Immediately following surgery.
  The patient's cooperation during the surgery period was graded by the surgeon choosing a number on a scale from one to ten considering 1 as totally cooperative (calm and steady fixing) and 10 as totally uncooperative (marked eye and head movement and/or lid squeezing).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, MD, Principal Investigator — Assiut University
Locations (1):
- Tiba Eye Center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramirez DA, Brodie FL, Rose-Nussbaumer J, Ramanathan S. Anxiety in patients undergoing cataract surgery: a pre- and postoperative comparison. Clin Ophthalmol. 2017 Nov 10;11:1979-1986. doi: 10.2147/OPTH.S146135. eCollection 2017. PMID 29184388